CLINICAL TRIAL: NCT00280969
Title: Open-label Randomized Multicenter Study of Once Daily Antiretroviral Treatment Regimen Comparing Ritonavir Boosted Atazanavir to Efavirenz
Brief Title: Comparing the Effectiveness Between Ritonavir Boosted Atazanavir and Efavirenz for the First HIV Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Medical Center of Japan (Other Government)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Shinichi Oka, M.D., Director general, AIDS Clinical Center, International Medical Center of Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QD001
Record Dates: First submitted 2006-01-22; First posted 2006-01-24 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection
Keywords: HIV infection; treatment; efavirenz; atazanavir; ritonavir
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atazanavir arm (Experimental): Patients are treated with ritonavir 100mg boosted atazanavir 300mg along with Epzicom.
  Interventions: Drug: atazanavir arm
- efavirenz arm (Active Comparator): Patients are treated with efavirenz 300mg along with Epzicom.
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: atazanavir arm — Patients are treated with ritonavir 100mg boosted atazanavir 300mg along with Epzicom.
  Arms: atazanavir arm
Drug: efavirenz — Patients are treated with efavirenz 300mg along with Epzicom.
  Arms: efavirenz arm

SUMMARY:
A selection study in treatment naive HIV patients to compare the virologic success rate of once daily antiretroviral treatment regimens at the 48th week with Epzicom(lamivudine and abacavir) plus efavirenz and Epzicom plus ritonavir boosted atazanavir. The superior regimen will be hired to the comparative study to the current first line regimen (tenofovir plus lamivudine plus efavirenz)

DETAILED DESCRIPTION:
A selection study in treatment naive HIV patients to compare the virologic success rate of once daily antiretroviral treatment regimens at the 48th week with Epzicom(lamivudine and abacavir) plus efavirenz and Epzicom plus ritonavir boosted atazanavir. The superior regimen will be hired to the comparative study to the current first line regimen (tenofovir plus lamivudine plus efavirenz)

The primary endpoint is antiretroviral effect at the 48th week.

The secondary endpoint is;1. Evaluation of immunological effect and safety in 48 weeks. 2.Evaluation of antiretroviral effect, immunological effect and safety in 49 to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* serological diagnosis of HIV infection
* male aged over 20 years old
* CD4 at enrollment between 100 to 300
* body weight over 40kg
* enable to obtain the written informed consent

Exclusion Criteria:

* Patients who are considered unable to complete 48 weeks of study by their physician.
* Patients who have gastrointestinal symptom which may interfere the absorption of antiretrovirals, or have swallowing problems.
* Patients who have the history of hypersensitivity with lamivudine.
* Hepatitis B carrier.
* Blood test results within 4 weeks prior to the randomization; hemoglobin less than 9g/dl, platelet less than 50,000/mm3, neutrophils less than 1000/mm3, serum total bilirubin more than 2.0mg/dl, GOT/GPT/LDH more than two times of upper normal limit, serum creatinine more than 1.2mg/dl.
* Patients who have had radiation or chemotherapy within 4 weeks prior to the randomization or will have the treatment during the study .
* Patients who have had immunomodulating agent such as systemic use of corticosteroid or interferon within 4 weeks prior to the randomization. Inhaled corticosteroid is the exception.
* Patients who have diabetes, congestive heart failure, cardiomyopathy, or other serious medical condition.
* Patients with AIDS defining illness.
* Patients with known resistant strains to efavirenz, atazanavir, ritonavir, lamivudine and abacavir prior to the study.
* Patients with acute retroviral syndrome.
* Patients with psychiatric disorder.
* Patients whose physician consider the study enrollment inappropriate.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Antiretroviral effect at the 48th week | 48 weeks

SECONDARY OUTCOMES:
1. Evaluation of immunological effect and safety in 48 weeks. | 48 weeks
2.Evaluation of antiretroviral effect, immunological effect and safety in 49 to 96 weeks. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Oka, M.D., phD., Study Chair — International Medical Center of Japan
Locations (1):
- International Medical Center of Japan, Shinjuku, Tokyo, Japan

REFERENCES:
- [Result] Honda M, Ishisaka M, Ishizuka N, Kimura S, Oka S; Japanese Anti-HIV-1 QD Therapy Study Group. Open-label randomized multicenter selection study of once daily antiretroviral treatment regimen comparing ritonavir-boosted atazanavir to efavirenz with fixed-dose abacavir and lamivudine. Intern Med. 2011;50(7):699-705. doi: 10.2169/internalmedicine.50.4572. Epub 2011 Apr 1. PMID 21467701